CLINICAL TRIAL: NCT07115797
Title: Anterior Repositioning Splint With or Without Arthrocentesis and Platelet-rich Plasma Injection In TMD Patients With Anterior Disc Displacement With Reduction: A Randomized Controlled Clinical Trial
Brief Title: ARS vs ARS With Arthrocentesis and PRP Injection in DDWR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Saleh Thabit Ali, Master's candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARS+- PRP & Arthrocentesis
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: TMJ Disc Displacement With Reduction; TMD; PRP Injection
Keywords: ARS-PRP-Arthrocentsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the observers will be blind to which group this case belongs. evaluators, and statisticians will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): ARS
  Interventions: Other: ARS
- intervention (Active Comparator): arthrocentesis then PRP injection and then ARS
  Interventions: Other: arthrocentesis - PRP injection -ARS

INTERVENTIONS:
Other: arthrocentesis - PRP injection -ARS — oarthrocentesis then PRP injection and then ARS
  Arms: intervention
Other: ARS — Insertion Of ARS Only
  Arms: Comparator

SUMMARY:
This study will be conducted to assess the effect of anterior repositioning splint and arthrocentesis with platelet-rich plasma injection compared to anterior repositioning splint only, in TMD patients with anterior disc displacement with reduction

DETAILED DESCRIPTION:
Anterior repositioning splint (ARS) allows the mandible to assume an anterior position to centric occlusion, providing a more favorable condyle-disc relationship in the fossa so that normal function can be established. The goal is to eliminate the signs and symptoms associated with disc-interference disorders. Maintaining the mandible in a temporary therapeutic position in which click is eliminated and thereby allowing the disc to reposition

A study by (Mohamed & Abd el Azizi, 2021) Found that ARS showed a significant reduction of pain and increase in maximum mouth opening after 1 month and an increase in MMO. Platelet-rich plasma (PRP) is a therapeutic agent consisting essentially of a platelet concentrate and associated growth factors taken and centrifuged from a sample of the patient's blood. It was initially introduced in the fields of stomatology, maxillofacial/plastic surgery, and reconstructive surgery in the 1990s and its clinical use is due to its potential healing properties through cell recruitment, proliferation, differentiation, and consequently, tissue remodeling. It has been found to have several advantages over the use of corticosteroids in the treatment of TMJ degenerative and inflammatory conditions, the most remarkable being its lack of serious and/or irreversible adverse effects. Treatment with PRP injections has reported anti-inflammatory, analgesic and antibacterial properties and, at the same time, restores intra-articular levels of hyaluronic acid, increases glycosaminoglycan chondrocyte synthesis, balances joint angiogenesis, and induces stem cell migration.

Explanation for choice of comparators:

Anterior repositioning splint (ARS) therapy is a common conservative method for treating disc-displacement-related (TMDs). ARS can be fixed on the maxilla or mandible and it usually maintains the protrusion status through an anterior guidance ramp The protrusion of the mandible changes the disc condyle relationship and is widely used in intra-articular TMD treatment. This method can significantly improve pain symptoms. Thus, it can also be used in pain-related TMDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from internal derangement anterior disc displacement
* Mouth Opening: Limited range of motion or difficulty with full mouth opening
* Symptoms: Patients who report typical symptoms of TMJ dysfunction, such as pain, discomfort, or clicking sounds in the joint, especially when opening or closing the mouth.
* Clicking: Audible clicking.
* Pain: Pain or tenderness around the TMJ, often radiating to the ear, temple, or neck.

Exclusion Criteria:

* Blood dyscrasias and Uncontrolled systemic diseases.
* Rheumatoid Arthritis.
* Infection in the pre-auricular area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Maximum pain-free interincisal opening measured in mm by caliper | from enrollment to the end of study at 6 months

SECONDARY OUTCOMES:
Pain measured by VAS scale | from enrollment to the end of study at 6 months